CLINICAL TRIAL: NCT05544851
Title: The Effect of the Education Provided to Reproductive Age Women on the Prevention of Sexually Transmitted Diseases With the Teach Beck Method on Their Behaviors
Brief Title: The Effect of Education Given to Reproductive Age Women by Teach Back Method on Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Mustafa KILAVUZ, Principal investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: HASANKAU; FERİDE YİĞİT (Other: HASANKU)
Record Dates: First submitted 2021-12-07; First posted 2022-09-19 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Sexually Transmitted Diseases
Keywords: reproductive age; Sexually Transmitted Disease; Women Health
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Inclusion Criteria / Patient
  Women of reproductive age (range 18-49 years) No history of STD, literate, Ability to understand and answer questions Those who have not received training on STDs before,
  Exclusion Criteria from Research
  Getting training on STDs before Absence from education for at least two sessions, Women with a history of STD (HIV, HPV, etc.) disease will be excluded from the study.
Who Masked: Participant
Masking Description: Inclusion Criteria / Patient
  Women of reproductive age (range 18-49 years) No history of STD, literate, Ability to understand and answer questions Those who have not received training on STDs before,
  Exclusion Criteria from Research
  Getting training on STDs before Absence from education for at least two sessions, Women with a history of STD (HIV, HPV, etc.) disease will be excluded from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educated Reproductive Women (Experimental): Inclusion Criteria / Patient
  Women of reproductive age (range 18-49 years) No history of STD, literate, Ability to understand and answer questions Those who have not received training on STDs before,
  Exclusion Criteria from Research
  Getting training on STDs before Absence from education for at least two sessions, Women with a history of STD (HIV, HPV, etc.) disease will be excluded from the study.
  Interventions: Other: Education
- Non-Educated Reproductive Women (Experimental): Inclusion Criteria / Patient
  Women of reproductive age (range 18-49 years) No history of STD, literate, Ability to understand and answer questions Those who have not received training on STDs before,
  Exclusion Criteria from Research
  Getting training on STDs before Absence from education for at least two sessions, Women with a history of STD (HIV, HPV, etc.) disease will be excluded from the study.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Participants who meet the sample selection criteria will be informed about the scope of the study and their verbal and written consent will be obtained. Women who met the sample selection criteria and were accepted into the study group will be randomly assigned to the intervention and control groups. Personal Information Form, "Behaviors for Protection from Sexually Transmitted Diseases Scale" will be applied to the participants in the intervention and control groups.

SUMMARY:
Sexually transmitted infections (STIs) are an important public health problem as they affect more than 1 million people worldwide every day. The extent of sexually transmitted diseases is still unknown due to underreporting, underdiagnosis or asymptomatic course of these diseases. When the literature is examined, it is seen that the incidence of STD has increased in recent years. The prevalence of premarital sexual intercourse as a result of the decrease in the age of sexual maturity but the increase in the age at marriage in general plays an important role in this increase. It is estimated that 46.8 million of 450 million people in the 15-49 age group living in the European region, including Turkey, have treatable STIs. STD can lead to many serious health problems such as infertility, ectopic pregnancy, cancer, chronic pelvic pain, pelvic adhesions and even death. Moreover, eye diseases, central nervous system infection and death may occur in the baby of an infected mother. In the report of the "Study on Sexual and Reproductive Health in Young People" conducted in Turkey in 2007, it was determined that young people do not have sufficient information about the reproductive organs, structure and physiology, health problems that may arise due to STD, HIV/AIDS, and ways of protection (6).An effective education; can significantly affect the quality of care, personal safety and satisfaction. One of the most effective and successful methods used in education is the Teach-Back method. Tell What You've Learned is a communication and education method used in health education for patients to remember and understand important information about diagnosis, treatment, medications or care. Tell What You've Learned is explained as a method that can be easily used for almost any interaction between healthcare team members and patients and can strengthen team understanding. It is recommended that all personnel, not only clinical caregivers, should use the method effectively in the health care system. It is stated that the conceptual framework of this method is based on the individuals receiving health services to present the information by arranging them according to themselves. It is considered as an effective method in terms of determining whether the transferred information is understood correctly.

It is stated that 40-80% of the individuals who consult or immediately forget the information given to them about their health. Various factors that cause communication problems between healthcare professionals and clients during information transfer affect the clarity and permanence of the information given.The "Tell What You Have Learned" method is also expressed as closing the loop, and it is reported to be an effective method when used to eliminate the communication gap between healthcare professionals and service recipients. In addition, it is stated that the use of the method to control the materials (educational brochure, training guide, etc.) used by individuals leaving the hospital to access health information will have a positive effect on health outcomes. From another point of view; It is predicted that it will increase the health literacy rate, and it is accepted as a research-based health literacy intervention that enriches the communication between the health care provider and the service recipient, improves the health outcomes of the individual.

DETAILED DESCRIPTION:
Purpose of the research; The aim of this study is to examine the effects of the education given to women of reproductive age to protect themselves from sexually transmitted diseases on their behaviors.

Research Hypotheses

1. Education made with "Tell What You Have Learned" method positively affects women's prevention behaviors from STD.
2. Is the Scale of Behavior for Protection from Sexually Transmitted Diseases a valid scale?
3. Is the Scale of Behavior for Protection from Sexually Transmitted Diseases a reliable scale? Importance of Research I. Although the prevalence of sexually transmitted diseases is high, it is stated in the literature that there is a lack of information on this subject in the society. This study, which is planned to be carried out, aims to develop women's behaviors towards prevention of STD, to recognize the symptoms in the early stages of the disease and to treat them in a short time. The study aimed to protect women from STD.

It is important in terms of developing a new scale as well as increasing their awareness and improving their behaviors.

II. The results of the study, it is planned to contribute to the development of community health by increasing the STD awareness and health promotion behaviors of women of reproductive age for protection from STD.

Research Questions

1. Does the education made with the "Tell What You Have Learned" method have an effect on the prevention behaviors from STD?
2. Is the Scale of Behavior for Protection from Sexually Transmitted Diseases a valid and reliable scale?

Ethical Aspect of Research:

The research will be carried out by Hasan Kalyoncu University Ethics Committee Presidency and Istinye University Bahçelievler Medical Park Ethics Committee Presidency with the permission of the ethics committee.

Application permission will be obtained from İstinye University Bahçelievler Medical Park hospital where the research will be conducted.

Within the scope of the research, the confidentiality of the patients' name and information will be taken as a basis.

No fee will be requested from the patients for their participation in the research and no additional fee will be paid to the patients who accept the research.

Participation in the research will be done on a voluntary basis. Participants who want to leave the study will be excluded from the study.

Type and Time of Research:

The research was planned methodologically and experimentally. As a methodological study, "Behavioral Scale for Protection from Sexually Transmitted Diseases" will be developed. Experimentally given to women of reproductive age with the "Tell What You Learned" method for protection from sexually transmitted diseases.

The effect of education on behavior will be investigated. The research will be carried out between May 2022 and October 2022.

Population and Sample of the Research The universe of the research; Between May 2022 and October 2022, women of reproductive age who applied to Bahçelievler Medical Park Hospital, Gynecology Outpatient Clinic will be formed.

Sample of the research:

The sample of the first stage of the research; determined by the number of items in the scale. When the literature is reviewed, it is seen that the number of items will be 5-10 times as many participants and factor analysis will be applied in the data.

It is seen that the sample size should be at least 50. The sample will be determined according to the number in the item pool.

In the calculation of the sample size of the second stage of the study, the data of the study titled "The Effect of Breastfeeding Education Given by Tell What You've Learned Method on Breastfeeding Success: Randomized Controlled Study" were used (8). Alpha margin of error is 5%, research power is 80% (Effect Size: 0.80) It was determined that there should be at least 26 people in each group. Since there may be losses during the follow-ups, a total of 70 women will be included in the sample, including at least 35 intervention groups and at least 35 control groups.

Location and Characteristics of the Research The research will be carried out at the İstinye University Bahçelievler Medikalpark Hospital, Obstetrics and Gynecology Polyclinic, affiliated to the Istanbul Health Directorate.

I Data Collection Tools Data will be collected using the "Personal Information Collection Form", "Behavior Scale for Protection from Sexually Transmitted Diseases" and "Tell Me What You Have Learned" observation tool. Personal Information Form: personal information form developed by the researcher in line with the literature; Demographic characteristics of women (age, employment status, etc.), Questions about Sexual Health (and It consists of questions categorized under the headings. The personal information form will be finalized by taking the opinion of the academicians specialized in the field of Midwifery and Obstetrics and Gynecology Nursing.

Behavior Scale for Protection from Sexually Transmitted Diseases: It will be used after the scale is developed by the researcher and the validity and reliability studies are completed.

Tell What You've Learned Observation Tool: To evaluate the observations of the practitioner using the Teach-Back method by monitoring the method of application by a competent person.

For this purpose, it is recommended to evaluate by using the "Teach-Back Observation Tool". It is based on observing whether the method is applied correctly by a competent person. It is aimed to use the method effectively and to eliminate the deficiencies by observing the skill level of the practitioner regarding the method. The Turkish adaptation of the Tell What You Have Learned Observation Tool was done by Kul Uçtu. Evaluation of the application of the "Tell What You Have Learned" method in this study, At every stage of the research, the "Tell What You Have Learned" Observation Tool will be used.

Statistical Analysis of Data

The data will be evaluated using the SPSS 22.0 statistical package program. The construct validity of the scale will be examined using the SPSS AMOS program. Sample adequacy will be determined by Kaiser-Meyer-Olkin (KMO) analysis, the suitability of the sample for factor analysis will be determined by Barlett's Test analysis, and explanatory and confirmatory factor analysis will be performed. Internal consistency of the scale, Cronbach's Alpha coefficient, the effect of each item on the total score, item-total correlation coefficients, whether the scale is an additive scale or not. Tukey will be determined by a splicability test. The final form of the scale will be created from the items with the highest reliability.

Tests planned to be used in the analysis of the data, Single Sample Kolmogorov Smirnov Test for examining the conformity of numerical variables with normal distribution, Student's t test for comparing quantitative variables with normal distribution among women, and comparing non-normally distributed quantitative variables.

Mann Whitney U test and Chi-square test will be used to compare categorical data.

ELIGIBILITY:
Inclusion Criteria for Research

* Women of reproductive age (range 18-49 years)
* No history of STD, literate,
* Ability to understand and answer questions
* Those who have not received training on STDs before,

Exclusion Criteria from Research

* Getting training on STDs before
* Absence from education for at least two sessions,
* Women with a history of STD (HIV, HPV, etc.) disease will be excluded from the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Reproductive women between 18-49
Enrollment: 1000 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
The importance of education | 12 months
  Data collection stages:
  Participants who meet the sample selection criteria will be informed about the scope of the study and their verbal and written consent will be obtained. Women who met the sample selection criteria and were accepted into the study group will be randomly assigned to the intervention and control groups. Personal Information Form, "Behaviors for Protection from Sexually Transmitted Diseases Scale" will be applied to the participants in the intervention and control groups. HTA training will be applied to the intervention group with the tell what you learned method, and clinical routines will be applied to the control group. The maximum score to be taken from the scale is 105, the minimum score is 21.The scale used scores the behaviors of the participants. Participants with low scores have deficiencies in behaviors towards protection from sexually transmitted diseases. After the training is given to the participants, their repetitive behavior will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Feride Yiğit, Study Director — Hasan Kalyoncu Unıvercıty
Locations (1):
- Hasan Kalyoncu Unıvercıty, Gaziantep, Turkey (Türkiye)